CLINICAL TRIAL: NCT04989894
Title: Investigating the Quality of Recovery After Childbirth
Brief Title: Quality of Recovery After Childbirth
Status: Recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Sng Ban Leong, Head of Department, Women's Anaesthesia, KK Women's and Children's Hospital
Other Study IDs: 2021/2160
Record Dates: First submitted 2021-07-04; First posted 2021-08-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Quality of Life; Childbirth; Maternal Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this proposed study, the investigators hope to assess the quality of recovery after delivery in a local population that would take into account physiological and psychological parameters to better understand the recovery process after delivery. The investigators will identify risk factors, especially those that are modifiable and associated with a poorer ObsQoR score and hence a poor quality of recovery after delivery. This data may then be used to educate women and manage expectations in the postpartum period, and help develop potential therapeutic interventions.

DETAILED DESCRIPTION:
Traditional postpartum outcome measures do not describe the patient experience or quality of recovery (QoR) after childbirth. A recent obstetric-specific recovery tool (ObsQoR-10) has been developed to assess the quality of recovery in patients in various mode of delivery on aspects of pain, drug side effects, comfort, control, ability to hold and feed the baby, independent mobilization and achievement of personal hygiene. However, this questionnaire is not yet validated in Asian population, especially in Chinese- and Malay-speaking patients.

The investigators aim to investigate the validity, reliability, feasibility, and responsiveness of the Chinese and Malay translated versions of ObsQoR-10. The investigators will first perform a pre-test in 5-10 patients for each language, of which an interview will be conducted to seek for their feedback and suggestions. Modification of questionnaire will be done if necessary, followed by recruitment of 112 patients at postpartum day 1 to fill in the Chinese/Malay translated ObsQoR-10 and other questionnaires related to their mood, anxiety and pain. In this proposed study, the investigators hope to assess the quality of recovery after delivery in a local population that would take into account physiological and psychological parameters to better understand the recovery process after delivery. The investigators will identify risk factors, especially those that are modifiable and associated with a poorer ObsQoR score and hence a poor quality of recovery after delivery. This data may then be used to educate women and manage expectations in the postpartum period, and help develop potential therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-50 years old;
* Able to read and understand written Chinese;
* Primiparous and having singleton pregnancy;
* Delivered via spontaneous vaginal delivery, or elective cesarean delivery;
* ≥38 gestational week.

Exclusion Criteria:

* Failed neuraxial analgesia in those receiving elective cesarean delivery;
* General anaesthesia;
* Intrapartum cesarean delivery;
* Women whose infants have died;
* Mother or baby requiring ICU after delivery;
* Assisted/ operative vaginal delivery.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only parturients who have given birth will be recruited.
Study Population: Only parturients who have given birth will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of ObsQoR-10-Chinese after 60 mins | Postpartum day 1; 1 day
  Repeat of ObsQoR-10-Chinese at 60 mins after the first postpartum day 1 ObsQoR-10-Chinese and its correlation to the previous hour ObsQoR-10-Chinese (test-retest reliability)
Change of ObsQoR-10-Malay after 60 mins | Postpartum day 1; 1 day
  Repeat of ObsQoR-10-Malay at 60 mins after the first postpartum day 1 ObsQoR-10-Malay and its correlation to the previous hour ObsQoR-10-Malay (test-retest reliability)

SECONDARY OUTCOMES:
Correlation between ObsQoR-10-Chinese and global health status | Postpartum day 1; 1 day
  Correlation of postpartum day 1 ObsQoR-10-Chinese scores with EQ-5D-3L-Chinese scores and global health Visual analog scale (VAS) (GHVAS; how good or bad is patient's health today, in her opinion, from 100 'Best imaginable health state' to 0 'Worst imaginable health state')
Correlation between ObsQoR-10-Malay and global health status | Postpartum day 1; 1 day
  Correlation of postpartum day 1 ObsQoR-10-Malay scores with EQ-5D-3L-Malay scores and global health Visual analog scale (VAS) (GHVAS; how good or bad is patient's health today, in her opinion, from 100 'Best imaginable health state' to 0 'Worst imaginable health state')
Correlation between ObsQoR-10-Chinese and recovery | Postpartum day 1; 1 day
  Correlation of postpartum day 1 ObsQoR-10-Chinese scores with good recovery (postpartum 1 GHVAS >=70mm) vs poor recovery (postpartum day 1 GHVAS < 70mm)
Correlation between ObsQoR-10-Malay and recovery | Postpartum day 1; 1 day
  Correlation of postpartum day 1 ObsQoR-10-Malay scores with good recovery (postpartum 1 GHVAS >=70mm) vs poor recovery (postpartum day 1 GHVAS < 70mm)
Correlation between ObsQoR-10 and length of hospital stay | Postpartum day 1; 1 day
  Correlation of postpartum day 1 ObsQoR-10 scores with length of hospital stay (time from delivery to discharge)
Correlation between ObsQoR-10 and acute pain scores | Postpartum day 1; 1 day
  Correlation of postpartum day 1 ObsQoR-10 scores with acute pain scores (numerical rating scale 0 to 10; 0 being no pain and 10 being the pain worst imaginable)
Correlation between ObsQoR-10 and breastfeeding self-efficacy | Postpartum day 7; 1 day
  Correlation of postpartum day 1 ObsQoR-10 scores with breastfeeding self-efficacy measured by breastfeeding self-efficacy scale- short form (BSES-SF). Breastfeeding self-efficacy refers to a mother's confidence and perception of how well she can breastfeed her infant. The 14-item self-administered BSES-SF comes in a 5-point Likert-type scale where 1 indicates not at all confident and 5 indicates always confident. Scores are summed to produce a range from 14 to 70, with higher scores indicating higher levels of breastfeeding self-efficacy.
Correlation between ObsQoR-10 and postnatal depressive symptoms | Postpartum day 7; 1 day
  Correlation of postpartum day 1 ObsQoR-10 scores with postnatal depressive symptoms measured by Edinburgh Postnatal Depression Scale (EPDS). Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self reporting scale to evaluate the postnatal depression. Participants are asked to respond according to how they have felt in the past seven days. Each item is measured on a 4-point scale (0-3), with a total score in the range of 0 to 30. A higher total score indicates a greater degree of depressive symptoms. A score of 10 and above indicates clinically significant depressive symptoms.
Time on the use of ObsQoR-10 | Postpartum day 1; 1 day
  Time taken in minutes to complete the ObsQoR-10 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, Principal Investigator — Head and Senior Consultant, Women's Anaesthesia
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tan HS, Tan CW, Sultana R, Yang L, Mok MUS, Sng BL. The correlation between quality of recovery and parturient outcomes after Cesarean delivery: a cohort study. Can J Anaesth. 2024 Sep;71(9):1272-1281. doi: 10.1007/s12630-024-02799-x. Epub 2024 Aug 12. PMID 39134784